CLINICAL TRIAL: NCT03337750
Title: An Open-Trial of Web-Prolonged Exposure (Web-PE) Among Active-Duty Military
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Texas (Other); VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carmen McLean, Adjunct Assistant Professor, University of Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20170600H
Record Dates: First submitted 2017-11-03; First posted 2017-11-09 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Posttraumatic Stress Disorder; Combat Disorders
Keywords: Combat; Psychological Treatment; Military; Psychotherapy; Trauma; Posttraumatic Stress; Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders; Wounds and Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Web-PE (Experimental): Ten 60-minute psychotherapy sessions over 8 weeks, focused on gradually confronting distressing trauma-related memories and reminders. Web-PE is an internet-based version of prolonged exposure (PE) for posttraumatic stress disorder (PTSD).
  Interventions: Behavioral: Web-PE Therapy

INTERVENTIONS:
Behavioral: Web-PE Therapy — Ten 60-minute psychotherapy sessions over 8 weeks, focused on gradually confronting distressing trauma-related memories and reminders. Web-PE is an internet-based version of prolonged exposure (PE) for posttraumatic stress disorder (PTSD).
  Other Names: Internet-based prolonged exposure

SUMMARY:
It is urgent to make evidence-based treatments (EBTs) for military personnel readily accessible in order to meet the growing demand for effective and efficient treatment for posttraumatic stress disorder (PTSD) in a timely manner. Effective EBTs for PTSD are available, but barriers to accessing care can deter military personnel from receiving treatment. Web-treatments represent an innovative way to overcome these barriers. The efficacy of previously developed web-treatments for PTSD appear promising, however, they are not based on treatment protocols with strong empirical support for their efficacy. No study to date has examined web-treatment of PTSD using a well-established treatment program.

The purpose of this open trial is to examine the efficacy of 10 sessions of a web-version of Prolonged Exposure (PE), "Web-PE," delivered over 8-weeks in 40 active-duty military personnel and veterans with PTSD who deployed post 9-11. Up to 60 individuals will be consented to obtain data from 40 for analysis. Participants will be assessed at pre-treatment and 1- and 3-months after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Active-duty military personnel and veterans who have deployed post 9/11
* Seeking treatment for PTSD
* Significant PTSD symptoms as determined by a PCL-5 score greater than or equal to 31
* Has experienced a Criterion A event that is a specific combat-related event or high magnitude operational experience that occurred during a period of recent military deployment
* Able to speak and read English and access to an internet-connected computer
* Indication that the participant plans to be able to participant in the study for the next three months following the first assessment

Exclusion Criteria:

* Diagnosis of bipolar disorder or psychotic disorder, as determined by participant self-report)
* Current substance dependence, as determined by participant self-report)
* Diagnosis of a moderate or severe traumatic brain injury, as determined by participant self-report)
* Current suicidal ideation severe enough to warrant immediate attention, as determined by participant self-report)
* Currently engaged in evidence-based treatment for PTSD (e.g. Prolonged Exposure Therapy or Cognitive Processing Therapy), as determined by participant self-report.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
PTSD CheckList-5 (PCL-5) | Change from baseline to 1-month follow-up (post-treatment)
  A 20-item self-report measure of PTSD symptoms as defined by the DSM-5. Higher scores indicate greater PTSD symptom severity.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Change from baseline to 1-month follow-up (post-treatment)
  A 9-item measure of the severity of depressive symptoms. Higher scores indicated greater depressive symptom severity.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Center for the Treatment and Study of Anxiety, University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- See also: Study enrollment page — https://studypages.com/s/are-you-a-veteran-or-service-member-dealing-with-posttraumatic-stress-participate-in-a-web-based-treatment-study-357599/
- See also: STRONG STAR consortium — https://tango.uthscsa.edu/strongstar/